CLINICAL TRIAL: NCT01785628
Title: The Impact of Pharmacological and Electric Modulation of NMDA Pathway on the Cognitive Flexibility and Volitional Movement Preparation in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chon-Haw Tsai, The Chief, Department of Neurology, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DMR98-IRB-296
Record Dates: First submitted 2011-06-24; First posted 2013-02-07 (Estimated); Results first posted 2013-08-22 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Parkinson's Disease With Dementia
Keywords: Parkinson's disease; dementia; NMDA; event related potential; Bereitschaftspotential
MeSH Terms: conditions — Parkinson Disease; Dementia | interventions — Sarcosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sarcosine capsule (Experimental): Oral capsules of Sarcosine (0.5g capsule) 1g / bid for 8 weeks.
  Interventions: Dietary Supplement: Sarcosine Capsule
- Placebo capsule (Placebo Comparator): Oral capsules of Placebo (Dextrin 0.5g capsule) 1g / bid for 8 weeks.
  Interventions: Dietary Supplement: Placebo Capsule

INTERVENTIONS:
Dietary Supplement: Sarcosine Capsule — Sarcosine is a glycine transporter-1 (GlyT-1) inhibitor. By blocking glycine uptake, sarcosine increases synaptic glycine concentration to enhance NMDA receptor function.
  Arms: Sarcosine capsule
Dietary Supplement: Placebo Capsule — Placebo is dextrin composition.
  Arms: Placebo capsule

SUMMARY:
The project will investigate the effect of pharmacological and electric modulation of N-methyl-D-aspartate (NMDA) pathway on the cognitive flexibility and volitional movement preparation in patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
Sarcosine (also called N-methylglycine) is an endogenous GlyT-1 inhibitor. By blocking glycine uptake, sarcosine increases synaptic glycine concentration to enhance NMDA receptor function. NMDA receptor, a subtype of ionotropic glutamate receptors, serves important functions in the brain, including learning, memory, cognition, and neural plasticity under physiological conditions and contributes to neurodegeneration in pathophysiological processes. NMDA receptor represents collectively a group of heteromeric tetramers. Every NMDA receptor is a protein complex, typically composed of two NR1 subunits and two NR2 subunits that together form the NMDA receptor ion channel. It requires two receptor agonists (glutamate for the NR2 binding site and glycine for the NR1 binding site) to open the ion channel for NMDA receptor activation. Clinically, modulation through the NMDA-NR1-glycine site is preferred to avoid the excitotoxicity associated with the glutamate site activation.8 In addition, recent animal studies have shown that dopamine secretion can be enhanced by either blocking the striatal NR2 or by activation of the NMDA-receptor glycine site. In the project, we will focus on pharmacological enhancement of NMDA-glycine receptor function based on increasing synaptic glycine concentration by sarcosine administration to examine whether enhancing NMDA-glycine receptor activity can improve the neuropsychiatric symptoms, cognition and hopefully motor function in PD-D patients

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of PD-D will be based on the criteria proposed by 2007 movement disorders PD-D task force. (Emre M et.al. Mov Disord 2007; 22:1689-1707)

Exclusion Criteria:

* Acute confusion due to systemic illnesses or drug intoxication.
* Major depression
* Features compatible with "Probable Vascular dementia.
* Patient who is pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chon-Haw Tsai, MD, PHD, Principal Investigator — Department of Neurology, China Medical University Hospital, Taichung, Taiwan
Locations (1):
- China Medical University Hospital/Neuro Depart., Taichung, Taiwan

REFERENCES:
- [Derived] Tsai CH, Huang HC, Liu BL, Li CI, Lu MK, Chen X, Tsai MC, Yang YW, Lane HY. Activation of N-methyl-D-aspartate receptor glycine site temporally ameliorates neuropsychiatric symptoms of Parkinson's disease with dementia. Psychiatry Clin Neurosci. 2014 Sep;68(9):692-700. doi: 10.1111/pcn.12175. Epub 2014 Apr 14. PMID 24612097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of recruitment period: 05-Aug-2010 to 08-Jun-2012 Type of location: Hospital, Medical China Universities, Neurology clinic.
Pre-assignment Details: The diagnosis of PD-D was based on the criteria proposed by 2007 movement disorders PD-D task force. 30 patients were enrolled.
Period: Overall Study
Arm/Group | Sarcosine Capsule | Placebo Capsule
Started | 15 | 15
Completed | 13 | 12
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sarcosine Capsule | Placebo Capsule | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 14 | 15 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 76.3 (5.3) | 77.3 (6.6) | 76.8 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 8 | 11 | 19
Region of Enrollment [Number; unit: participants]
  Taiwan | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) From Baseline to 8 Weeks.
Description: Outcome is defined as change in total Unified Parkinson's Disease Rating Scale (UPDRS) between the baseline to 8 weeks. The UPDRS score has three parts, part I (Mentation, Behavior and Mood), Part II (Activities of Daily Living) and Part III (Motor Examination). Each consisting of questions answered on a 0-4 point scale. The minimum total score possible is 0 and the maximum total score possible is 176. Higher scores indicating more severe symptoms.
Time Frame: baseline to 8 weeks.
Population: The Intent-to-Treat (ITT) Population comprised all randomised patients who took at least one dose of study medication or placebo and who had a valid baseline efficacy measure and at least one post-baseline efficacy measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sarcosine Capsule | Placebo Capsule
Number analyzed (Participants) | 15 | 15
Scores on a scale
  baseline | 71.6 (21.8) | 66.7 (23.1)
  V1(2-week) | 67.9 (20.9) | 65.2 (24)
  V2(4-week) | 69.3 (22.5) | 67.6 (22.4)
  V3(8-week) | 71.3 (25.1) | 68.3 (21.7)

2. Secondary Outcome: Change in Cognitive Abilities Screening Instrument (CASI) From Baseline to 8 Weeks.
Description: The Cognitive Abilities Screening Instrument (CASI) has a score range of 0 to 100 and provides quantitative assessment on attention, concentration, orientation, short-term memory, long-term memory, language abilities, visual construction, list-generating fluency, abstraction, and judgment. With a higher score indicating Symptom improvement.
Time Frame: baseline to 8 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sarcosine Capsule | Placebo Capsule
Number analyzed (Participants) | 15 | 15
Scores on a scale
  Baseline | 50.9 (23.8) | 63.9 (23.9)
  V2(4 weeks) | 53.1 (21.8) | 63.9 (22.5)
  V3(8weeks) | 52.4 (24.0) | 63.9 (24.6)

3. Secondary Outcome: Change in Clinical Dementia Rating (CDR) From Baseline to 8 Weeks.
Description: The CDR is a 5-point scale used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care. With a higher score indicating more severe symptoms.
Time Frame: baseline to 8 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sarcosine Capsule | Placebo Capsule
Number analyzed (Participants) | 15 | 15
Scores on a scale
  Baseline | 2.3 (2.1) | 1.1 (1.2)
  V2(4 weeks) | 2.1 (2.0) | 1.1 (1.3)
  V3(8 weeks) | 2.0 (2.1) | 1.1 (1.3)

4. Secondary Outcome: Change in Neuropsychiatry Inventory (NPI) From Baseline to 8 Weeks.
Description: The NPI scale has 12 domains: delusions, hallucinations, agitation, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor behavior, night-time behavior disturbances, and appetite and eating abnormalities. The total score ranges from 0 to 144, where the score for a domain is defined as the product of frequency (range: 1-4) and severity (range: 1-3). Each domain has a maximum score of 12 and with a higher score indicating more severe symptoms.
Time Frame: baseline to 8 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sarcosine Capsule | Placebo Capsule
Number analyzed (Participants) | 15 | 15
Scores on a scale
  Baseline | 18.4 (13.4) | 14.9 (11.2)
  V1(2weeks) | 14.8 (13.3) | 14.1 (11.9)
  V2(4 weeks) | 12.4 (13.9) | 11.7 (11.6)
  V3(8 weeks) | 18.1 (13.6) | 13.3 (10.4)

5. Secondary Outcome: Change in Behavioral Pathology in Alzheimer's Disease Rating Scale (Behave-AD) From Baseline to 8 Weeks.
Description: The Behave-AD includes the assessment of symptoms and a global rating of caregiver distress. A total of 25 symptoms in 7 clusters are rated: paranoid and delusional ideation, hallucinations, aggressiveness, activity disturbances, diurnal rhythm disturbances, affective disturbances and anxieties, and phobias. Caregivers rate behavioral symptoms over the preceding 2 weeks on a 0 to 3 scale. The caregiver also determines a global assessment of caregiver distress on a scale of 0 to 3. The maximum score is 75 and with a higher score indicating more severe symptoms.
Time Frame: baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sarcosine Capsule | Placebo Capsule
Number analyzed (Participants) | 15 | 15
Scores on a scale
  Baseline | 10.0 (7.6) | 7.9 (6.5)
  V1(2 weeks) | 8.4 (7.9) | 5.2 (4.7)
  V2(4 weeks) | 7.5 (8.1) | 6.8 (6.8)
  V3(8 weeks) | 9.4 (8.8) | 6.4 (6.9)

6. Secondary Outcome: Change in Hamilton Depression Rating Scale (HAM-D) From Baseline to 8 Weeks.
Description: The HAM-D is a 21-item rating scaled which includes an emphasis on behavioral symptoms and somatic complaints that neglects self-reported feelings of distress; and an intermingling of frequency and intensity of symptoms. The total score ranges from 0 to 64: ten items are ranked on a scale from 0 to 4; 9 items are ranked 0 to 2; and 2 items are ranked 0 to 3. With a higher score indicating more severe symptoms.
Time Frame: baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sarcosine Capsule | Placebo Capsule
Number analyzed (Participants) | 15 | 15
Scores on a scale
  Baseline | 11.8 (8.0) | 7.6 (3.5)
  V1(2 weeks) | 9.9 (7.7) | 7.6 (2.4)
  V2(4 weeks) | 10.1 (7.6) | 7.8 (3.9)
  V3(8 weeks) | 11.0 (7.4) | 7.3 (3.2)

7. Secondary Outcome: Change in Beck Depression Inventory-II (BDI-II) From Baseline to 8 Weeks.
Description: The BDI-II is a 21-item self-report questionnaire assessing the current severity of depression symptoms. Each item is scored on a scale of 0 to 3 and the total score ranges from 0 to 63. With a higher score indicating more severe symptoms.
Time Frame: baseline to 8 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sarcosine Capsule | Placebo Capsule
Number analyzed (Participants) | 15 | 15
Scores on a scale
  Baseline | 14.3 (10.1) | 9.9 (4.2)
  V1(2 weeks) | 15.6 (9.7) | 10.5 (5.2)
  V2(4 weeks) | 15.8 (11.2) | 10.2 (4.6)
  V3(8 weeks) | 17.5 (11.7) | 9.8 (5.7)

8. Secondary Outcome: Change in The 39-item Parkinson's Disease Questionnaire (PDQ-39) From Baseline to 8 Weeks.
Description: The PDQ-39 contains 39-items covering 8 discrete dimensions: mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, and bodily discomfort. Each question is scored on a 5-point scale and recoded to 0 to 4 for the analysis. The total score can range from 0 to 132 and with a higher score indicating more severe symptoms.
Time Frame: baseline to 8 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sarcosine Capsule | Placebo Capsule
Number analyzed (Participants) | 15 | 15
Scores on a scale
  Baseline | 68.0 (28.2) | 64.8 (19.5)
  V1(2 weeks) | 67.9 (29.3) | 60.9 (18.9)
  V2(4 weeks) | 65.9 (26.4) | 60.9 (17.5)
  V3(8 weeks) | 63.7 (28.9) | 60.1 (18.2)

9. Other Pre Specified Outcome: Change in Brain Imaging by 18F-FDG PET From Baseline to 8 Weeks.
Description: 18F-FDG PET scan : 8 patients for treatment and placebo groups,respectively.
Time Frame: baseline to 8 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Brain Imaging by [99mTc]TRODAT-1 From Baseline to 8 Weeks.
Description: [99mTc]TRODAT-1 : 7 patients for treatment and placebo groups, respectively.
Time Frame: baseline to 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Sarcosine Capsule | Placebo Capsule
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sarcosine Capsule (N=15) | Placebo Capsule (N=15)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes